CLINICAL TRIAL: NCT00826098
Title: Platelet Rich Plasma (PRP) in Total Knee Replacement: A Prospective, Randomized, Single-blind, Single-center Clinical Study to Evaluate the Effect of Platelet Rich Plasma (PRP) on Short-term Patient Outcomes Following Total Knee Replacement
Brief Title: Platelet Rich Plasma (PRP) in Total Knee Replacement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Exactech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR07-004
Record Dates: First submitted 2009-01-20; First posted 2009-01-21 (Estimated); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Osteoarthritis; Inflammatory Arthritis
Keywords: Total knee replacement; Platelet Rich Plasma; PRP; Biologic; Randomized
MeSH Terms: conditions — Osteoarthritis; Arthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (PRP) (Experimental): Total knee replacement with PRP
  Interventions: Biological: Platelet Rich Plasma
- 2 (non-PRP) (No Intervention): Total knee replacement without PRP

INTERVENTIONS:
Biological: Platelet Rich Plasma — Addition of PRP to total knee replacement procedure
  Other Names: Accelerate PRP
  Arms: 1 (PRP)

SUMMARY:
Clinical study to evaluate the effect of platelet rich plasma (PRP), a derivative of a patient's whole blood, on short-term patient outcomes following total knee replacement (TKR).

DETAILED DESCRIPTION:
The purpose of this clinical study is to evaluate the effect of platelet rich plasma (PRP), a derivative of a patient's whole blood, on short-term patient outcomes following total knee replacement (TKR). The hypothesis is that change in short-term hemoglobin (Hgb) levels is less dramatic in patients who undergo TKR with the addition of PRP when compared to patients who undergo TKR without PRP.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is a male or female who is undergoing primary unilateral surgery or the first surgery of a staged bilateral total knee replacement where the second stage will be at least 6 weeks later PRP in Total Knee.
2. Patient agrees to be blinded to their treatment group assignment.
3. Patient is willing and able to return for follow-up over at least a six (6) week post-operative period although longer follow-up is desired
4. Patient agrees to participate by signing an IRB approved Informed Consent Form

Exclusion Criteria:

1. Patient will have a staged bilateral total knee replacement with the second stage to be performed less than 6 weeks after the first stage surgery
2. Patient has had previous surgery on the operative knee that will necessitate the removal of existing hardware (e.g. previous osteotomy)
3. Patient has a known adverse reaction or sensitivity to bovine (cow) thrombin (used as part of the platelet rich plasma system) or other bovine-derived products
4. Patient has hemoglobin < 12.0 (males), < 11.0 (females)
5. Patient clinically significant anxiety disorder
6. Patient is on therapeutic anticoagulation medication and has an INR > 1.3
7. Patient has a severe bleeding disorder
8. Patient has a known addiction to drugs or alcohol, including, but not limited to: chronic daily use of narcotic medications for more than 90 days prior to surgery
9. Patient is pregnant
10. Patient is a prisoner
11. Patient is involved in a personal litigation (e.g. Worker's Compensation) that relates to their knee surgery
12. Patient is actively participating in an investigational medical device, drug, or biologic clinical trial (active defined as having treatment within the last 30 days)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-12; Primary Completion 2011-06 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Hemoglobin level | Change in hemoglobin (Hgb) level (preop compared to postop day 2)
  Hemoglobin level analysis

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Moody, MD, Principal Investigator — Central Maine Orthopaedics, PA; Pasquale Petrera, MD, Principal Investigator — Peninsula Orthopedic Associates
Locations (2):
- United States (2):
  - Center for Joint Replacement, St. Mary's Regional Medical Center, Lewiston, Maine
  - Peninsula Orthopedic Associates, Salisbury, Maryland